CLINICAL TRIAL: NCT02871141
Title: Effects of Electroconvulsive Therapy on Neuronal, Immunological and Hormonal Parameters in Patients With Affective Disorders
Brief Title: Multimodal Imaging of ECT Effects
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Simone Grimm, PD Dr.rer.nat. Simone Grimm, Charite University, Berlin, Germany
Other Study IDs: BA 3578_ECT
Record Dates: First submitted 2016-08-09; First posted 2016-08-18 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Electroconvulsive Therapy; Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ECT group: Patients with a major depressive episode treated with ECT. Patients will be investigated (i) prior to the 1st ECT session, (ii) after the 4th ECT session, (iii) after the 12th ECT session, and (iv) 6 months after the 1st ECT session.
  Interventions: Procedure: electroconvulsive therapy
- Antidepressant group: Patients with a major depressive episode treated with antidepressants. Patients will be investigated (i) prior to treatment, (ii) after 10 days of treatment, (iii) after 4 weeks of treatment, and (iv) after 6 months.
  Interventions: Drug: Antidepressant

INTERVENTIONS:
Procedure: electroconvulsive therapy — electroconvulsive therapy
  Groups: ECT group
Drug: Antidepressant — Antidepressant
  Groups: Antidepressant group

SUMMARY:
The project aims to investigate markers of neural activity and connectivity, neurochemistry, hypothalamic-pituitary-adrenal (HPA) axis activity, inflammation and neuronal plasticity underlying treatment response and remission after ECT. These measures will be assessed in depressive patients prior, during and after ECT and also after 6 months. Furthermore, we will investigate a control group of depressive patients treated with antidepressants.

DETAILED DESCRIPTION:
About 30% of patients suffering from major depressive disorder (MDD) do not respond sufficiently to established pharmacological, psychotherapeutic, or somatic treatment. Treatment-resistant MDD is associated with illness chronicity, a reduced quality of life, and a higher risk for suicide. For these patients, electroconvulsive therapy (ECT) is a well-established treatment strategy with response rates of 60% to 80%, making it the most potent and rapidly acting treatment for MDD. Despite the frequent and widespread use of ECT for more than 70 years, the exact neurobiological mechanisms underlying its efficacy remain unclear. In a broader sense, understanding the therapeutic effects of ECT may also shed some more light on the pathophysiological causes of severe depression and the mechanisms of action of an effective treatment. Eventually, the elucidation of the effects of ECT could allow for their reproduction in a less invasive way and with a more benign side-effect profile, thereby resulting in an significantly enhanced treatment of MDD. To achieve this, though, we need first to understand better how ECT influences brain function. The proposed project therefore aims to investigate markers of neural activity and connectivity, neurochemistry, HPA axis activity, inflammation and neuronal plasticity underlying treatment response and remission after ECT. These measures will be assessed in depressive patients prior, during and after ECT and also after 6 months. Furthermore, we will investigate a control group of depressive patients treated with antidepressants. This treatment-specific approach will enable us to disentangle which behavioral, neuronal, hormonal and immunological alterations are crucial for an antidepressant response and might be used for response prediction. More generally, the project will greatly broaden our understanding of the mechanisms underlying the profound antidepressant effect of ECT and thereby shed some more light on the pathophysiological causes of MDD and the mechanisms of action of an effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* current diagnosis of Major Depression
* severity of current symptoms on a clinical level as indicated by scores of the Hamilton Scale of Depression
* age 25 to 60 in order to exclude cases of late-onset depression and age- associated changes in brain functions and volume
* right handedness
* fluency in spoken and written German
* treatment resistant depression, i.e. at least with two failed antidepressant treatment trials as assessed with the Antidepressant Treatment History Form (ATHF)

Exclusion Criteria:

* history of psychosis or mania, current eating disorder, obsessive- compulsive disorder (OCD), current self-harm, current substance abuse or dependence
* history of traumatic brain injury
* current treatment with glutamate- modulating medication.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Depressive patients from a primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in functional connectivity between medial and lateral prefrontal regions | 4 timepoints (ECT group: prior to 1st ECT, after the 4th ECT, after the 12th ECT, after 6 months; antidepressant group: prior to treatment, after 10 days, after 4 weeks , after 6 months
  Patients in the ECT group will be investigated (i) prior to the 1st ECT session, (ii) after the 4th ECT session, (iii) after the 12th ECT session, and (iv) 6 months after the 1st ECT session. Patients in the antidepressant group will be investigated (i) prior to treatment, (ii) after 10 days of treatment, (iii) after 4 weeks of treatment, and (iv) after 6 months. Measurements will be conducted using functional magnetic resonance imaging.
Changes in functional activity in medial and lateral prefrontal regions | 4 timepoints (ECT group: prior to 1st ECT, after the 4th ECT, after the 12th ECT, after 6 months; antidepressant group: prior to treatment, after 10 days, after 4 weeks , after 6 months
  Patients in the ECT group will be investigated (i) prior to the 1st ECT session, (ii) after the 4th ECT session, (iii) after the 12th ECT session, and (iv) 6 months after the 1st ECT session. Patients in the antidepressant group will be investigated (i) prior to treatment, (ii) after 10 days of treatment, (iii) after 4 weeks of treatment, and (iv) after 6 months. Measurements will be conducted using functional magnetic resonance imaging.
Changes in neurotransmitter concentrations in medial and lateral prefrontal regions | 4 timepoints (ECT group: prior to 1st ECT, after the 4th ECT, after the 12th ECT, after 6 months; antidepressant group: prior to treatment, after 10 days, after 4 weeks , after 6 months
  Patients in the ECT group will be investigated (i) prior to the 1st ECT session, (ii) after the 4th ECT session, (iii) after the 12th ECT session, and (iv) 6 months after the 1st ECT session. Patients in the antidepressant group will be investigated (i) prior to treatment, (ii) after 10 days of treatment, (iii) after 4 weeks of treatment, and (iv) after 6 months. Measurements will be conducted using functional magnetic resonance spectroscopy.
Changes in levels of cytokines, cortisol and BDNF | 4 timepoints (ECT group: prior to 1st ECT, after the 4th ECT, after the 12th ECT, after 6 months; antidepressant group: prior to treatment, after 10 days, after 4 weeks , after 6 months
  Patients in the ECT group will be investigated (i) prior to the 1st ECT session, (ii) after the 4th ECT session, (iii) after the 12th ECT session, and (iv) 6 months after the 1st ECT session. Patients in the antidepressant group will be investigated (i) prior to treatment, (ii) after 10 days of treatment, (iii) after 4 weeks of treatment, and (iv) after 6 months. Serum (BDNF, cytokines) and plasma (cortisol) levels will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Malek Bajbouj, MD, Principal Investigator — Charité
Locations (1):
- Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gruzman R, Hempel M, Domke AK, Hartling C, Stippl A, Carstens L, Bajbouj M, Gartner M, Grimm S. Investigating the impact of rumination and adverse childhood experiences on resting-state neural activity and connectivity in depression. J Affect Disord. 2024 Aug 1;358:283-291. doi: 10.1016/j.jad.2024.02.068. Epub 2024 Feb 20. PMID 38387672